CLINICAL TRIAL: NCT01917721
Title: Phase 2 Study to Assess the Efficacy and Safety of Doxycycline in Preventing Coronary Artery Aneurysm Formation and Progression
Brief Title: Doxycycline Treatment to Prevent Progressive Coronary Artery Dilation in Children With Kawasaki Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Responsible Party: Principal Investigator, Andras Bratincsak, MD, PhD, Clinical Assistant Professor, Hawaii Pacific Health
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-005
Record Dates: First submitted 2013-04-26; First posted 2013-08-07 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Kawasaki Disease; Coronary Aneurysm
Keywords: Kawasaki disease; doxycycline; coronary artery aneurysm
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — Doxycycline; Immunoglobulins, Intravenous; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Experimental): These patients will receive doxycycline at the acute phase of their disease
  Interventions: Drug: Doxycycline
- Placebo (Active Comparator): The comparative arm of the study will receive standard care and placebo for Kawasaki disease, but not doxycycline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — The interventional arm of the study will receive doxycycline 4.4 mg/kg/day for 21 days besides receiveing standard care: IVIG and/or Remicade.
  Arms: Doxycycline
Drug: Placebo — Standard medical care and placebo will be provided to the comparative arm of the study administering IVIG and/or Remicade, but not doxycycline.
  Other Names: IVIG and Remicade
  Arms: Placebo

SUMMARY:
Kawasaki disease (KD) affects infants and young children causing inflammation of the skin and blood vessels including the coronary arteries of the heart. Despite the currently available therapy, about one third of children develop enlargement of the coronary arteries that can lead to serious complications such as coronary artery stenosis, heart attack and even death.

Kawasaki disease is the most common heart disease in children in the USA and it is especially common among the children of Hawaii. Every year, 50-90 children are diagnosed with KD in Hawaii and unfortunately there is no medication available to successfully prevent coronary artery damage in a subset of cases.

During the first few weeks of the illness, cells of the immune system attack the coronary arteries and release a special substance (MMP) that is responsible for the coronary artery enlargement. There is a common antibiotic, doxycycline that can specifically block the action of this special substance (MMP). Research done on animals with KD showed that doxycycline was able to block this special substance and prevent enlargement of coronary arteries. Research in adults with enlargement of the main artery in their abdomen also showed that doxycycline may improve the outcome. Based on these studies doxycycline may be a promising therapy for children with KD, who develop enlargement of the coronary arteries.

The investigators' proposed research study will assess the usefulness of doxycycline in preventing the progressive enlargement of coronary arteries in children with KD. The investigators plan to perform a small (pilot) study to evaluate how good is doxycycline in preventing coronary artery enlargement. The investigators will treat 50 children with KD and enlarged coronary arteries for three weeks with doxycycline and assess the change in coronary arteries as well as the blood levels of the special substance (MMP). If doxycycline proves to be beneficial in this small study, the investigators are going to design a large research study involving multiple institutions on Hawaii and the mainland and will recruit more children to be certain about the value of the proposed treatment. The investigators' proposal may change the treatment protocol of KD and could present a possible treatment for children with enlarged coronary arteries preventing potentially devastating consequences.

DETAILED DESCRIPTION:
This research study attempts to reveal whether coronary artery dilation in patients with Kawasaki disease refractory to standard therapy could be prevented using a matrix metalloproteinase inhibitor: doxycycline.

Hypothesis The investigators hypothesize that oral administration of doxycycline for two weeks during the acute phase of Kawasaki disease (KD) effectively blocks matrix metalloproteinase-9 (MMP-9) activity in the coronary arteries and therefore prevents the progression of coronary artery dilation and aneurysm formation in children with KD.

Rationale There is no specific treatment for children with KD, who develop coronary artery dilation or aneurysm. Based on the animal studies and adult trials showing beneficial effect of doxycycline on coronary artery dilation and abdominal aneurysms, this selective MMP-9 inhibitor offers a promising therapeutic strategy to prevent progressive coronary artery dilation in children with KD.

Specific aims

1. Measure serum MMP-9 activity, tissue inhibitor of metalloproteinase 1 activity (TIMP-1), serum levels of degradation products due to MMP-9 activity (elastin and gelatin degradation products) before and after treatment with doxycycline in children with KD.
2. Compare serum MMP-9 activity and degradation product levels of children receiving only standard therapy for KD (IVIG, infliximab) with children receiving standard therapy and doxycycline treatment.
3. Measure the coronary artery diameters before and after doxycycline treatment in children with KD.
4. Compare coronary artery measurements of children receiving only standard therapy for KD (IVIG, infliximab) with children receiving standard therapy and doxycycline treatment.
5. Design a multi-center prospective randomized blinded placebo-controlled trial to assess the efficacy of doxycycline in preventing coronary artery dilation and aneurysm.

ELIGIBILITY:
Inclusion Criteria:

Treatment arm: Patients aged 1 month to 21 years with confirmed KD will be included in the study if they meet the following criteria:

1. Patients with dilation of the right or left anterior descending coronary artery beyond a z-score of +2.5 during the acute febrile phase of KD.
2. Patients with aneurysms of the right or left main coronary arteries during the acute febrile phase of KD.
3. Patients with refractory KD after initial treatment with IVIG and dilated coronary arteries on an echocardiogram during the first month of KD.

Comparison arm: Patients aged 1 month to 18 years with confirmed KD, who do not meet inclusion criteria to be included in the treatment group.

1.Patients with right or left anterior descending coronary artery measurements below a z-score of +2.5 during the acute febrile phase of KD.

Exclusion Criteria:

The following patients will be excluded from this study:

1. Patients with clinically incomplete KD.
2. Patients whose parents refuse to administer doxycycline.
3. Patients with acute renal failure.
4. Patients with chronic liver and kidney disease.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Coronary artery diameter change | 24 months
  We will assess the change (+ or -) of coronary artery diameter from the beginning of doxycycline administration to the end of doxycycline administration and for an additional 2 months beyond that.

SECONDARY OUTCOMES:
Assess the change in MMP-9 level | 24 months
  We will draw blood samples before, during and after the administration of doxycyline to assess the effect on MMP-9 (matrix metalloproteinase 9).
Assess a change in TIMP level | 24 months
  We will draw blood samples before, during and after the administration of doxycyline to assess the effect on MMP-9 (matrix metalloproteinase 9) and TIMP (tissue inhibitor of matrix metalloproteinase).

CONTACTS AND LOCATIONS:
Overall Officials: Andras Bratincsak, MD PhD, Principal Investigator — Hawaii Pacific Health
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bratincsak A, Limm-Chan BN, Nerurkar VR, Ching LL, Reddy VD, Lim E, Shohet RV, Melish ME. Study design and rationale to assess Doxycycline Efficacy in preventing coronary Artery Lesions in children with Kawasaki disease (DEAL trial) - A phase II clinical trial. Contemp Clin Trials. 2018 Feb;65:33-38. doi: 10.1016/j.cct.2017.11.014. Epub 2017 Dec 5. PMID 29313803